CLINICAL TRIAL: NCT06931314
Title: The Impact of Muscle Energy Technique and Aromatherapy on Pain, Disability and Sleep Quality in Office Workers With Nonspecific Neck Pain
Brief Title: The Impact of Muscle Energy Technique and Aromatherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayça Aytar (Other)
Responsible Party: Sponsor-Investigator, Ayça Aytar, doçent, Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA24/57
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain
Keywords: Lavender Oil; İsometric Contraction; aromatherapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: The people who will be included in our study will be examined in 3 groups: Muscle energy technique (MET), aromatherapy and control group.
  People in the manual energy technique and aromatherapy group will be given an application for 4 weeks in addition to exercise, while the control group will be given only exercise.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Muscle energy technique (MET) Group (Active Comparator): The MET group will be given an average of 20 minutes of exercise, 2 days a week for 4 weeks. The muscle energy technique (post isometric relaxation technique) for the upper trapezius and levator scapula muscles will be applied for 3 to 5 repetitions, using 20% of the maximum isometric contraction for 7 to 10 seconds, holding the stretch beyond the resistance barrier for 30 to 60 seconds. Since these muscles are overactive due to muscle imbalances, they will be determined as target muscles. The total treatment period is 4 weeks and 8 sessions.
  Interventions: Procedure: Muscle Energy Technique
- Aromatherapy Group (Active Comparator): The aromatherapy group will also receive an application 2 days a week for 4 weeks. A 20-minute lavender oil message will be applied to the neck area (with Euploraj and Petrisaj techniques). All aromatherapy interventions will be performed at 23°C. Essential oils will be purchased from a certified organic and tested company and will be used diluted. The application will be applied to the participants in the face-down position, with the arms in the inverted T position for 15 minutes. The application will be applied twice a week for 4 weeks.
  Interventions: Procedure: Aromatherapy massage
- Control Group (No Intervention): The patients in the control group will be given exercises in the form of a home program consisting of neck isometric, posture and stretching exercises by the physiotherapist. The exercises will start with stretching exercises and continue with neck isometric exercises in a way that does not cause pain. The participants will be asked to do the exercises twice a day, every day of the week for 4 weeks, with 10 repetitions of each movement, and a brochure will be given about the exercises. Evaluation surveys will be applied at the end of the 0th and 4th weeks.

INTERVENTIONS:
Procedure: Aromatherapy massage — Aromatherapy massage refers to a massage to be performed on the neck area with lavender oil.
  Arms: Aromatherapy Group
Procedure: Muscle Energy Technique — Muscle Energy Technique is a form of manual therapy that uses active muscle contraction and relaxation to improve musculoskeletal mechanics and relieve pain.
  Arms: Muscle energy technique (MET) Group

SUMMARY:
Individuals with nonspecific neck pain who work at a desk will be included in the study. Individuals will be examined in 3 groups: Muscle energy technique (MET), aromatherapy and control group. All participants will be given home program-style exercises consisting of neck isometric, posture and stretching exercises by a physiotherapist. In addition to exercise, individuals in the MET and aromatherapy groups will be given exercises for 4 weeks, while the control group will be given only exercise. Evaluation questionnaires will be applied to participants at the end of the 0th and 4th weeks. At the end of the study, outcome measures between the groups and before and after data within the groups will be compared.

DETAILED DESCRIPTION:
Nonspecific neck pain (NSBP) can occur without any history of injury or specific pathology related to the musculoskeletal system, or as a result of a postural or mechanical cause. Studies conducted on office workers have shown that working at a desk for long periods of time causes significant pain in the neck region, although not primarily. There are many therapeutic modalities in the treatment of neck pain. However, manual therapy approaches have been increasingly popular in many countries in recent years. Muscle energy technique (MET) is a treatment approach that uses soft tissue or joint manipulation or mobilization to improve the musculoskeletal system and reduce pain, including stretching maneuvers after active muscle contraction and relaxation. The technique, defined as a type of massage application, is used by utilizing physiological properties such as viscoelastic properties of myofascial tissues. MET is among the physiotherapy methods that affect joint range of motion, spinal pain, tissue fluid drainage and proprioception. In the literature, in the study comparing the effects of MET and Thai massage treatment on neck pain, it was stated that their effects on pain were similar, but their effectiveness with different massages and aromatherapy was not investigated. Aromatherapy is another complementary treatment method used in the treatment of musculoskeletal system diseases. It is stated that the components of the essential oils used during aromatherapy massage reach the circulatory system through the lymph and blood vessels in the epidermis and affect the release of neurotransmitters such as dopamine, endorphin, noradrenaline and serotonin, thus reducing pain.Individuals with nonspecific neck pain who work at a desk will be included in the study. Individuals will be examined in 3 groups: Muscle energy technique (MET), aromatherapy and control group. All participants will be given home program-style exercises consisting of neck isometric, posture and stretching exercises by a physiotherapist. In addition to exercise, individuals in the MET and aromatherapy groups will be given exercises for 4 weeks, while the control group will be given only exercise. Evaluation questionnaires will be applied to participants at the end of the 0th and 4th weeks. At the end of the study, outcome measures between the groups and before and after data within the groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-55 years
* Female
* Office worker
* NP that has persisted for at least six months.

Exclusion Criteria:

* Individuals under the age of 18,
* Those with a history of neck-related surgery,
* Individuals with known serious pathologies (e.g., malignancy, inflammatory disorders, infection),
* Those with a history of trauma or fracture in the cervical spine,
* Individuals showing symptoms of cervical radiculopathy or myelopathy,
* Individuals known to have allergies to the oils to be used,
* Damaged skin,
* Individuals with a history of allergy to lavender and almond,
* Those with a history of respiratory system diseases,
* Individuals for whom massage and manipulation are contraindicated.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study involved 45 women diagnosed with nonspecific NP.
Enrollment: 45 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Neck Pain | The individuals participating in the study will be evaluated twice: before the application (week 0) and after the application (after 4 weeks).
  Visual Analog Scale (VAS) will be used to measure the pain intensity of the participants. It is evaluated by asking the individual to indicate the current situation they feel by drawing a line or a dot on the chart, on a straight line of ten centimeters, the two ends of which are defined by the parameter to be measured in the individual, and the pain intensity in the individual is calculated in this way.

SECONDARY OUTCOMES:
Neck Disability Index | The individuals participating in the study will be evaluated twice: before the application (week 0) and after the application (after 4 weeks).
  "Neck Disability Index (NDI) was used to assess the severity of neck disability (ND) in individuals participating in the study (Vernon & Mior, 1991; MacDermid et al., 2009). The index consists of 10 items including pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleep, and recreation. Participants rated the impact of neck pain by marking one of six boxes.
Pittsburgh Sleep Quality Index | The individuals participating in the study will be evaluated twice: before the application (week 0) and after the application (after 4 weeks).
  Pittsburgh Sleep Quality Index consists of seven subcomponents measuring subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction 26

CONTACTS AND LOCATIONS:
Overall Officials: Ayça AYTAR, Assoc.Prof., Study Director — Baskent University; Mustafa GÜLŞEN, Assoc.Prof., Study Chair — Baskent University; Selin ÖZEN, Assoc.Prof., Study Chair — Baskent University; Yasemin Kavuncubaşı Genç, Phd Cand, Study Chair — Baskent University; Aydan AYTAR, Professor, Study Director — University of Health Sciences Türkiye
Locations (1):
- Başkent University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phadke A, Bedekar N, Shyam A, Sancheti P. Effect of muscle energy technique and static stretching on pain and functional disability in patients with mechanical neck pain: A randomized controlled trial. Hong Kong Physiother J. 2016 Apr 14;35:5-11. doi: 10.1016/j.hkpj.2015.12.002. eCollection 2016 Dec. PMID 30931028
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Buttagat V, Muenpan K, Wiriyasakunphan W, Pomsuwan S, Kluayhomthong S, Areeudomwong P. A comparative study of Thai massage and muscle energy technique for chronic neck pain: A single-blinded randomized clinical trial. J Bodyw Mov Ther. 2021 Jul;27:647-653. doi: 10.1016/j.jbmt.2021.05.007. Epub 2021 May 11. PMID 34391301
- [Background] Canpolat M, Ortabağ T. Ofis Çalışanlarında Mobil Egzersizin Boyun Ağrısı Üzerine Etkisi. Istanbul Kent University Journal Of Health Sciences.2023;2(3): 22-25.
- [Background] Kanchanomai S, Janwantanakul P, Pensri P, Jiamjarasrangsi W. Risk factors for the onset and persistence of neck pain in undergraduate students: 1-year prospective cohort study. BMC Public Health. 2011 Jul 15;11:566. doi: 10.1186/1471-2458-11-566. PMID 21756362